CLINICAL TRIAL: NCT00567983
Title: Topical Cyclosporine and Disease Progression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Sanjay Rao, MD, Lakeside Eye Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13717A
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Disease Progression; Disease Severity; Staining; Schirmers; OSDI
MeSH Terms: conditions — Disease Progression | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1. (Active Comparator)
  Interventions: Drug: Restasis
- 2. (Placebo Comparator)
  Interventions: Drug: Endura

INTERVENTIONS:
Drug: Restasis — Restasis- (in the eye) Instill one drop twice daily Endura- (in the eye) Instill one drop twice daily
  Arms: 1.
Drug: Endura — Restasis- (in the eye) Instill one drop twice daily Endura- (in the eye) Instill one drop twice daily
  Arms: 2.

SUMMARY:
The purpose of this study is to evaluate the effect Restasis has in regards to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate dry eye symptoms

Exclusion Criteria:

* Current use of Restasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Disease Severity | 1 yr

SECONDARY OUTCOMES:
Staining | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rao, Principal Investigator — Lakeside Eye Clinic
Locations (1):
- Lakeside Eye Clinic, Chicago, Illinois, United States